CLINICAL TRIAL: NCT02130258
Title: Somatosensory Profiling in Radicular Pain Patients And it's Correlation With Treatment Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yi Zhang, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011P002234
Record Dates: First submitted 2014-04-24; First posted 2014-05-05 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Radiculopathy; Lower Extremity Radicular Pain
Keywords: Radicular; Pain; Epidural Steroid Injection
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- >30% Pain Relief (Other): All subjects have radicular pain and are scheduled to receive an epidural steroid injection (ESI) as a treatment. The ESI treatment is conducted by the subject's clinical physician and is not given as part of the research study procedures. Quantitative Sensory Testing (QST) will be conducted before and after the ESI treatment. QST consists of hot and cold temperature testing using the QST device. This group of subjects received greater than 30% pain relief.
  Interventions: Device: Quantitative Sensory Testing (QST); Procedure: Epidural Steroid Injection (ESI)
- <30% Pain Relief (Other): All subjects have radicular pain and are scheduled to receive an epidural steroid injection (ESI) as a treatment. The ESI treatment is conducted by the subject's clinical physician and is not given as part of the research study procedures. Quantitative Sensory Testing (QST) will be conducted before and after the ESI treatment. QST consists of hot and cold temperature testing using the QST device. This group of subjects received less than 30% pain relief.
  Interventions: Device: Quantitative Sensory Testing (QST); Procedure: Epidural Steroid Injection (ESI)

INTERVENTIONS:
Device: Quantitative Sensory Testing (QST) — Subjects will undergo hot and cold temperature testing using the QST device at two points: 1) Before ESI and 2) after ESI.
Procedure: Epidural Steroid Injection (ESI) — Subjects will receive an ESI by their clinical physician as part of their clinical treatment. This procedure is not given as part of the research study.

SUMMARY:
The investigators hypothesize that there may exist different quantitative sensory profiles between radicular pain patients who respond and those who do not respond to the standard therapy of epidural steroid injections (ESI).

DETAILED DESCRIPTION:
The investigators are comparing warm/cold sensation, heat/cold pain threshold, heat/cold pain tolerance, wind-up, and conditioned pain modulation (CPM) as measured by Quantitative Sensory Testing (QST) between subjects with a radicular pain condition. The investigators are comparing those who respond and those who do not respond to standard therapy (ESI) before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of lower extremity radicular pain regardless of specific or suspected etiologies
* scheduling an epidural steroid injection (ESI)

Exclusion Criteria:

* a major psychiatric disorder requiring a recent (within one month) hospitalization, such as major depression, bipolar disorder, schizophrenia, anxiety disorder, and psychosis
* subject is taking illicit or recreational drug detected through a urine toxicology screen
* subject has had an interventional pain management procedures within the last eight weeks that may alter QST responses including neuraxial or local anesthetic block
* subject had a change in dosage of neuromodulatory pain medication (including gabapentin, pregabalin, cymbalta, amitriptyline, nortriptyline, trileptal, etc) in the past two weeks
* subject is pregnant
* subject has pending litigation involving the current pain condition being treated and studied.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MGH Center for Translational Pain Research — http://www.massgeneral.org/translationalpainresearch/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from the MGH Center for Pain Medicine in Boston, MA.
Pre-assignment Details: 23 subjects were initially enrolled. 3 subjects were withdrawn before assignment to groups for the following reasons:
  1. sensory deficits at the site of QST and inability to complete questionnaires on own
  2. did not receive ESI which is a requirement for the study
Period: Overall Study
Arm/Group | >30% Pain Relief | <30% Pain Relief
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | >30% Pain Relief | <30% Pain Relief | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.55 (14.49) | 54.44 (11.56) | 56.15 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject was withdrawn before filling out questionnaires. Population description was not obtained.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 6 | 10 | 16
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 11 | 20
Opioid Use [Count of Participants; unit: Participants]
  Uses opioids | 1 | 6 | 7
  Does not use opioids | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Pre-epidural Warm Sensation Quantitative Sensory Testing (QST) Results
Description: QST tests for changes in spinal nerves. A small metal plate, called a thermode, is placed on the subject's arm. During the warm sensation test, the plate slowly increases in temperature.The subject will stop the test as soon as the plate feels warm. This temperature is recorded and can range from 32-53 degrees Celsius. The same test is repeated on the subject's leg that has radicular pain. The difference in temperatures from the test on the subject's arm and leg were analyzed.
Time Frame: Baseline measurement before the epidural injection
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | >30% Pain Relief | <30% Pain Relief
Number analyzed (Participants) | 9 | 11
Degrees Celsius | 2.68 (2.92) | 5.67 (3.22)
Statistical Analysis 1: Comparison: >30% Pain Relief vs <30% Pain Relief; Test type: Other; p = .04, Kruskal-Wallis

2. Primary Outcome: Post-epidural Continued Pain Modulation (CPM)
Description: CPM is a type of QST where the thermode is placed on the subject's non painful arm. Heat stimulation (47 degrees C, 4 seconds) was delivered to the thermode 4 times and the subject rated the pain felt by the heat stimulation on a visual analog scale (VAS) of 0-10. During the second heat stimulation, the subject immersed their hand (opposite from the arm with the thermode) in 12 degree C water and then rated the pain felt by the heat on a VAS of 0-10 (10 is the worst pain a subject can imagine, 0 is no pain). The final 2 heat stimuli were delivered (without using the hand submerged in water). This same test was repeated with the thermode on the subject's leg with radicular pain. The subject placed their hand contralateral to the painful leg in the cold water during the second heat stimulation. The VAS scores from each heat stimulation were averaged for the non-painful arm and the painful leg. The difference in averages between the arm and leg were then analyzed.
Time Frame: 4 weeks after the epidural injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | >30% Pain Relief | <30% Pain Relief
Number analyzed (Participants) | 9 | 11
units on a scale | -0.53 (2.01) | -4.08 (4.67)
Statistical Analysis 1: Comparison: >30% Pain Relief vs <30% Pain Relief; Test type: Other; p = .04, Kruskal-Wallis

3. Primary Outcome: Post-epidural Cold Pain Threshold QST Results
Description: The thermode is placed on the subject's arm. During the cold pain threshold test, the plate slowly decreases in temperature.The subject will stop the test when the plate is at their minimal tolerable temperature. This temperature is recorded and can range from 32-0 degrees Celsius. The same test is repeated on the subject's leg that has radicular pain. The difference in temperatures from the test on the subject's arm and leg were analyzed.
Time Frame: 4 weeks after the epidural injection
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | >30% Pain Relief | <30% Pain Relief
Number analyzed (Participants) | 9 | 11
Degrees Celsius | -0.60 (4.10) | -7.35 (9.11)
Statistical Analysis 1: Comparison: >30% Pain Relief vs <30% Pain Relief; Test type: Other; p = 0.04, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | >30% Pain Relief | <30% Pain Relief
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes